CLINICAL TRIAL: NCT06041256
Title: CLARA: A Phase 1/2 Multi-center, Randomized, Double-Masked, Prospective, Parallel-Arm Study of AURN001 in Subjects With Corneal Edema Secondary to Corneal Endothelial Dysfunction (ABA-1)
Brief Title: A Phase 1/2 Study of AURN001 in Subjects With Corneal Edema Secondary to Corneal Endothelial Dysfunction (ABA-1)
Acronym: CLARA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aurion Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABA-1
Record Dates: First submitted 2023-09-11; First posted 2023-09-18 (Actual); Results first posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Corneal Edema; Corneal Endothelial Dysfunction
MeSH Terms: conditions — Corneal Edema | interventions — Y 27632

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- AURN001 High (Experimental): Neltependocel High and Rho-associated protein kinase
  Interventions: Combination Product: AURN001
- AURN001 Medium (Experimental): Neltependocel Medium and Rho-associated protein kinase
  Interventions: Combination Product: AURN001
- AURN001 Low (Experimental): Neltependocel Low and Rho-associated protein kinase
  Interventions: Combination Product: AURN001
- Neltependocel (Experimental): Neltependocel - High
  Interventions: Biological: Corneal Endothelial Cells
- ROCK (Experimental): Rho-associated protein kinase (ROCK)
  Interventions: Drug: Y27632

INTERVENTIONS:
Combination Product: AURN001 — Corneal Endothelial Cells and Y27632
  Arms: AURN001 High; AURN001 Low; AURN001 Medium
Biological: Corneal Endothelial Cells — Corneal Endothelial Cells
  Arms: Neltependocel
Drug: Y27632 — Y27632
  Arms: ROCK

SUMMARY:
The goal of this clinical trial is to compare different doses of AURN001 in patients with corneal edema secondary to corneal endothelial dysfunction. The main questions the clinical trial aims to answer are whether AURN001 effective and safe. Participants will receive a single injection of AURN001. A comparison between low, medium, and high doses of AURN001 against the contribution of each element, cells alone and Y27632 alone, will be conducted to determine the effects on corneal edema.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of corneal edema secondary to corneal endothelial dysfunction, requiring surgery (full- or partial-thickness endothelial keratoplasty)
* BCVA between 65 Early Treatment of Diabetic Retinopathy Study (ETDRS) letters (i.e., 0.4 LogMAR or approximate 20/50 Snellen equivalent) and 5 ETDRS letters (i.e., 1.6 LogMAR or approximate 20/800 Snellen equivalent)

Exclusion Criteria:

* Have pre-operative corneal epithelial, sub-epithelial or stromal scarring or other opacity that is paracentral/central and visually significant, but not suspected to be secondary to corneal endothelial disease with the potential to improve from treatment in the study eye
* Have history or presence of an ocular disease other than corneal endothelial dysfunction that could affect vision or safety assessments

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2023-10-18 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2025-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Manager, OD, Study Director — Aurion Biotech
Locations (19):
- United States (16):
  - Aurion Biotech site, Little Rock, Arkansas
  - Aurion Biotech site, Los Angeles, California
  - Aurion Biotech site, San Francisco, California
  - Aurion Biotech site, Atlanta, Georgia
  - Aurion Biotech site, Indianapolis, Indiana
  - Aurion Biotech site, Wichita, Kansas
  - Aurion Biotech site, Minnetonka, Minnesota
  - Aurion Biotech site, Garden City, New York
  - Aurion Biotech site, Winston-Salem, North Carolina
  - Aurion Biotech site, Cincinnati, Ohio
  - Aurion Biotech site, Oklahoma City, Oklahoma
  - Aurion Biotech site, Bala-Cynwyd, Pennsylvania
  - Aurion Biotech site, Sioux Falls, South Dakota
  - Aurion Biotech site, Houston, Texas
  - Aurion Biotech site, Norfolk, Virginia
  - Aurion Biotech site, Seattle, Washington
- Canada (3):
  - Aurion Biotech site, Vancouver, British Columbia
  - Aurion Biotech site, Oakville, Ontario
  - Aurion Biotech site, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter, randomized, double-masked, parallel-arm, dose-ranging Phase 1/2 study evaluating safety, efficacy, and tolerability of AURN001 in participants with corneal edema due to endothelial dysfunction. Three dose levels were compared with neltependocel and Y-27632 alone to assess each component's contribution on efficacy and safety of AURN001.
Pre-assignment Details: A total of 97 participants were enrolled and received the study treatment.
Groups:
- Y-27632 100 µM: Participants received a single intracameral injection of Y-27632 (100 Micromolar [μM]) under local anesthesia.
- Neltependocel 1.0 × 10^6: Participants received a single intracameral injection of neltependocel 1.0 × 10^6 cells under local anesthesia.
- AURN001 (2.5 × 10^5 Neltependocel + Y-27632 100 µM): Participants received a single intracameral injection of neltependocel 2.5 × 10^5 cells administered with Y-27632 100 μM under local anesthesia.
- AURN001 (5.0 × 10^5 Neltependocel + Y-27632 100 µM): Participants received a single intracameral injection of neltependocel 5.0 × 10^5 cells administered with Y-27632 100 μM under local anesthesia.
- AURN001 (1.0 × 10^6 Neltependocel + Y-27632 100 µM): Participants received a single intracameral injection of neltependocel 1.0 × 10^6 cells administered with Y-27632 100 μM under local anesthesia.
Period: Overall Study
Arm/Group | Y-27632 100 µM | Neltependocel 1.0 × 10^6 | AURN001 (2.5 × 10^5 Neltependocel + Y-27632 100 µM) | AURN001 (5.0 × 10^5 Neltependocel + Y-27632 100 µM) | AURN001 (1.0 × 10^6 Neltependocel + Y-27632 100 µM)
Started | 21 | 18 | 19 | 19 | 20
Completed | 3 | 12 | 7 | 12 | 17
Not Completed | 18 | 6 | 12 | 7 | 3
Not completed — Withdrawal by Subject | 1 | 0 | 3 | 1 | 1
Not completed — Rescue | 17 | 6 | 9 | 6 | 2

BASELINE CHARACTERISTICS:
Population: Full Analysis Set comprised of all randomized participants who received any amount of study drug during intracameral injection.
Groups:
- Total: Total of all reporting groups
Arm/Group | Y-27632 100 µM | Neltependocel 1.0 × 10^6 | AURN001 (2.5 × 10^5 Neltependocel + Y-27632 100 µM) | AURN001 (5.0 × 10^5 Neltependocel + Y-27632 100 µM) | AURN001 (1.0 × 10^6 Neltependocel + Y-27632 100 µM) | Total
Number analyzed (Participants) | 21 | 18 | 19 | 19 | 20 | 97
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.3 (9.59) | 71.3 (9.93) | 74.7 (10.32) | 69.3 (6.91) | 71.6 (8.28) | 71.4 (9.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 10 | 5 | 15 | 55
  Male | 10 | 4 | 9 | 14 | 5 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 0 | 0 | 2
  Not Hispanic or Latino | 21 | 17 | 18 | 17 | 20 | 93
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 1 | 1 | 1 | 5
  White | 18 | 17 | 15 | 18 | 19 | 87
  More than one race | 0 | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving ≥15-letter Improvement in Best-corrected Visual Acuity (BCVA) at Month 6 - Imputed Data
Description: Best-corrected visual acuity was assessed using Early Treatment Diabetic Retinopathy Study(ETDRS) method, standard for vision testing. Standardized Sloan letter charts with 5 letters per line, decreasing by 0.1 logarithm of minimum angle of resolution (LogMAR) per line, were used at 4 meters (or 1 meter if ≤19 letters were read, with +0.75 spherical power added). Each correct letter equaled one point (0.02 LogMAR), with 85 letters (0.0 LogMAR) corresponding to 20/20 Snellen, 70 letters (+0.3) to 20/40, and 35 letters (+1.0) to 20/200. A gain of ≥15 letters (0.3 LogMAR, 3 lines) was clinically meaningful. Data from the study eye only were included in the analysis. Participants read letters aloud, guessing encouraged, and all responses recorded for accuracy. Data presented represent number of participants with available BCVA measurements at Month 6, with those who had missing data, underwent rescue surgery before Month 6, or discontinued study prior to Month 6 imputed as non-responders.
Time Frame: Month 6
Population: Full Analysis Set.
Measure: Number; unit: Percentage of participants
Groups:
- Neltependocel (1.0 × 10^6): Participants received a single intracameral injection of neltependocel 1.0 × 10^6 cells under local anesthesia.
Arm/Group | Y-27632 100 µM | Neltependocel (1.0 × 10^6) | AURN001 (2.5 × 10^5 Neltependocel + Y-27632 100 µM) | AURN001 (5.0 × 10^5 Neltependocel + Y-27632 100 µM) | AURN001 (1.0 × 10^6 Neltependocel + Y-27632 100 µM)
Number analyzed (Participants) | 21 | 18 | 19 | 19 | 20
Percentage of participants | 14.3 | 44.4 | 10.5 | 36.8 | 50.0
Statistical Analysis 1: Comparison: Y-27632 100 µM vs Neltependocel (1.0 × 10^6); Test type: Other; p = 0.0722, Fisher Exact; Difference in response rates = 30.2, 95% CI 2-sided [0.8 to 58.3]
Statistical Analysis 2: Comparison: Y-27632 100 µM vs AURN001 (2.5 × 10^5 Neltependocel + Y-27632 100 µM); Test type: Other; p > 0.9999, Fisher Exact; Difference in response rates = -3.8, 95% CI 2-sided [-28.1 to 20.6]
Statistical Analysis 3: Comparison: Y-27632 100 µM vs AURN001 (5.0 × 10^5 Neltependocel + Y-27632 100 µM); Test type: Other; p = 0.1482, Fisher Exact; Difference in response rates = 22.6, 95% CI 2-sided [-5.5 to 50.6]
Statistical Analysis 4: Comparison: Y-27632 100 µM vs AURN001 (1.0 × 10^6 Neltependocel + Y-27632 100 µM); Test type: Other; p = 0.0203, Fisher Exact; Difference in response rates = 35.7, 95% CI 2-sided [5.9 to 61.6]
Statistical Analysis 5: Comparison: Neltependocel (1.0 × 10^6) vs AURN001 (2.5 × 10^5 Neltependocel + Y-27632 100 µM); Test type: Other; p = 0.0293, Fisher Exact; Difference in response rates = -33.9, 95% CI 2-sided [-60.3 to -4.6]
Statistical Analysis 6: Comparison: Neltependocel (1.0 × 10^6) vs AURN001 (5.0 × 10^5 Neltependocel + Y-27632 100 µM); Test type: Other; p = 0.7431, Fisher Exact; Difference in response rates = -7.6, 95% CI 2-sided [-38.9 to 25.3]
Statistical Analysis 7: Comparison: Neltependocel (1.0 × 10^6) vs AURN001 (1.0 × 10^6 Neltependocel + Y-27632 100 µM); Test type: Other; p = 0.7568, Fisher Exact; Difference in response rates = 5.6, 95% CI 2-sided [-26.8 to 37.3]

2. Secondary Outcome: Change From Baseline in BCVA at Month 6
Description: Best-corrected visual acuity was assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) method, the standard for vision testing. Standardized Sloan letter charts with five letters per line, decreasing by 0.1 logarithm of the minimum angle of resolution (LogMAR) per line, were used at 4 meters (or 1 meter if ≤19 letters were read, with +0.75 spherical power added). Each correct letter equaled one point (0.02 LogMAR), with 85 letters (0.0 LogMAR) corresponding to 20/20 Snellen, 70 letters (+0.3) to 20/40, and 35 letters (+1.0) to 20/200. A gain of ≥15 letters (0.3 LogMAR, 3 lines) was clinically meaningful. Data from the study eye only were included in the analysis. Participants read letters aloud, guessing encouraged, and all responses recorded for accuracy. Baseline was defined as the last measurement prior to the study drug injection on Day 1. Change from baseline values was calculated as follow-up visit minus baseline visit.
Time Frame: Baseline (Day 1) and at Month 6
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: change in ETDRS letters
Arm/Group | Y-27632 100 µM | Neltependocel (1.0 × 10^6) | AURN001 (2.5 × 10^5 Neltependocel + Y-27632 100 µM) | AURN001 (5.0 × 10^5 Neltependocel + Y-27632 100 µM) | AURN001 (1.0 × 10^6 Neltependocel + Y-27632 100 µM)
Number analyzed (Participants) | 21 | 18 | 19 | 19 | 20
change in ETDRS letters | -25.5 (6.06) | -5.1 (6.41) | -15.7 (6.24) | -3.0 (6.25) | 10.4 (6.17)
Statistical Analysis 1: Comparison: Y-27632 100 µM vs Neltependocel (1.0 × 10^6); Test type: Other; p = 0.0232, ANCOVA; Least square mean difference = 20.4, 95% CI 2-sided [2.9 to 38.0]
Statistical Analysis 2: Comparison: Y-27632 100 µM vs AURN001 (2.5 × 10^5 Neltependocel + Y-27632 100 µM); Test type: Other; p = 0.2600, ANCOVA; Least square mean difference = 9.8, 95% CI 2-sided [-7.4 to 27.1]
Statistical Analysis 3: Comparison: Y-27632 100 µM vs AURN001 (5.0 × 10^5 Neltependocel + Y-27632 100 µM); Test type: Other; p = 0.0115, ANCOVA; Least square mean difference = 22.5, 95% CI 2-sided [5.2 to 39.9]
Statistical Analysis 4: Comparison: Y-27632 100 µM vs AURN001 (1.0 × 10^6 Neltependocel + Y-27632 100 µM); Test type: Other; p < 0.0001, ANCOVA; Least square mean difference = 36.0, 95% CI 2-sided [18.5 to 53.4]
Statistical Analysis 5: Comparison: Neltependocel (1.0 × 10^6) vs AURN001 (2.5 × 10^5 Neltependocel + Y-27632 100 µM); Test type: Other; p = 0.2403, ANCOVA; Least square mean difference = -10.6, 95% CI 2-sided [-28.4 to 7.2]
Statistical Analysis 6: Comparison: Neltependocel (1.0 × 10^6) vs AURN001 (5.0 × 10^5 Neltependocel + Y-27632 100 µM); Test type: Other; p = 0.8138, ANCOVA; Least square mean difference = 2.1, 95% CI 2-sided [-15.7 to 19.9]
Statistical Analysis 7: Comparison: Neltependocel (1.0 × 10^6) vs AURN001 (1.0 × 10^6 Neltependocel + Y-27632 100 µM); Test type: Other; p = 0.0834, ANCOVA; Least square mean difference = 15.5, 95% CI 2-sided [-2.1 to 33.2]

3. Secondary Outcome: Change From Baseline in Central Corneal Thickness (CCT) at Month 6
Description: Central corneal thickness was measured by pachymetry which is an essential anatomical marker for detecting the presence or absence of edema and serves as a supportive indicator of treatment efficacy. Baseline was defined as the last measurement prior to the study drug injection on Day 1. Change from baseline values was calculated as follow-up visit minus baseline visit.
Time Frame: Baseline (Day 1) and at Month 6
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: Microns
Arm/Group | Y-27632 100 µM | Neltependocel (1.0 × 10^6) | AURN001 (2.5 × 10^5 Neltependocel + Y-27632 100 µM) | AURN001 (5.0 × 10^5 Neltependocel + Y-27632 100 µM) | AURN001 (1.0 × 10^6 Neltependocel + Y-27632 100 µM)
Number analyzed (Participants) | 21 | 18 | 19 | 19 | 20
Microns | 67.5 (20.52) | -7.6 (22.17) | -13.8 (21.68) | -5.6 (21.91) | -14.2 (21.82)
Statistical Analysis 1: Comparison: Y-27632 100 µM vs Neltependocel (1.0 × 10^6); Test type: Other; p = 0.0147, ANCOVA; Least square mean difference = -75.1, 95% CI 2-sided [-135.2 to -15.1]
Statistical Analysis 2: Comparison: Y-27632 100 µM vs AURN001 (2.5 × 10^5 Neltependocel + Y-27632 100 µM); Test type: Other; p = 0.0077, ANCOVA; Least square mean difference = -81.3, 95% CI 2-sided [-140.5 to -22.0]
Statistical Analysis 3: Comparison: Y-27632 100 µM vs AURN001 (5.0 × 10^5 Neltependocel + Y-27632 100 µM); Test type: Other; p = 0.0165, ANCOVA; Least square mean difference = -73.1, 95% CI 2-sided [-132.6 to -13.7]
Statistical Analysis 4: Comparison: Y-27632 100 µM vs AURN001 (1.0 × 10^6 Neltependocel + Y-27632 100 µM); Test type: Other; p = 0.0079, ANCOVA; Least square mean difference = -81.7, 95% CI 2-sided [-141.4 to -22.0]
Statistical Analysis 5: Comparison: Neltependocel (1.0 × 10^6) vs AURN001 (2.5 × 10^5 Neltependocel + Y-27632 100 µM); Test type: Other; p = 0.8443, ANCOVA; Least square mean difference = -6.1, 95% CI 2-sided [-67.8 to 55.6]
Statistical Analysis 6: Comparison: Neltependocel (1.0 × 10^6) vs AURN001 (5.0 × 10^5 Neltependocel + Y-27632 100 µM); Test type: Other; p = 0.9490, ANCOVA; Least square mean difference = 2.0, 95% CI 2-sided [-60.1 to 64.1]
Statistical Analysis 7: Comparison: Neltependocel (1.0 × 10^6) vs AURN001 (1.0 × 10^6 Neltependocel + Y-27632 100 µM); Test type: Other; p = 0.8324, ANCOVA; Least square mean difference = -6.6, 95% CI 2-sided [-68.1 to 55.0]

4. Secondary Outcome: Percentage of Participants Achieving ≥15-letter Improvement in BCVA at All Timepoints - Observed Data
Description: Best-corrected visual acuity was assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) method, the standard for vision testing. Standardized Sloan letter charts with five letters per line, decreasing by 0.1 logarithm of the minimum angle of resolution (LogMAR) per line, were used at 4 meters (or 1 meter if ≤19 letters were read, with +0.75 spherical power added). Each correct letter equaled one point (0.02 LogMAR), with 85 letters (0.0 LogMAR) corresponding to 20/20 Snellen, 70 letters (+0.3) to 20/40, and 35 letters (+1.0) to 20/200. A gain of ≥15 letters (0.3 LogMAR, 3 lines) was clinically meaningful. Data from the study eye only were included in the analysis. Participants read letters aloud, guessing encouraged, and all responses recorded for accuracy. The data presented reflect only participants with non-missing BCVA at each corresponding visit.
Time Frame: At Week 4 and at Months 2, 3, 4.5, 6, 9 and 12
Population: Full Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Number; unit: percentage of participants
Arm/Group | Y-27632 100 µM | Neltependocel (1.0 × 10^6) | AURN001 (2.5 × 10^5 Neltependocel + Y-27632 100 µM) | AURN001 (5.0 × 10^5 Neltependocel + Y-27632 100 µM) | AURN001 (1.0 × 10^6 Neltependocel + Y-27632 100 µM)
Number analyzed (Participants) | 21 | 17 | 19 | 19 | 20
percentage of participants
  Week 4 | 4.8 | 5.9 | 10.5 | 5.3 | 10.0
  Month 2: number analyzed (Participants) | 6 | 6 | 7 | 8 | 10
  Month 2 | 0 | 16.7 | 0 | 0 | 10.0
  Month 3: number analyzed (Participants) | 15 | 17 | 17 | 19 | 19
  Month 3 | 6.7 | 35.3 | 11.8 | 21.1 | 26.3
  Month 4.5: number analyzed (Participants) | 12 | 14 | 14 | 17 | 19
  Month 4.5 | 0 | 42.9 | 14.3 | 29.4 | 36.8
  Month 6: number analyzed (Participants) | 6 | 14 | 12 | 16 | 19
  Month 6 | 50.0 | 57.1 | 16.7 | 43.8 | 52.6
  Month 9: number analyzed (Participants) | 3 | 12 | 8 | 13 | 18
  Month 9 | 33.3 | 58.3 | 37.5 | 38.5 | 50.0
  Month 12: number analyzed (Participants) | 3 | 12 | 7 | 12 | 17
  Month 12 | 0 | 58.3 | 28.6 | 66.7 | 76.5

5. Secondary Outcome: Change From Baseline in BCVA at All Other Timepoints
Description: as for outcome 2
Time Frame: Baseline (Day 1) and at Week 4, Months 2, 3, 4.5, 6, 9 and 12
Population: Full Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: change in ETDRS letters
Arm/Group | Y-27632 100 µM | Neltependocel (1.0 × 10^6) | AURN001 (2.5 × 10^5 Neltependocel + Y-27632 100 µM) | AURN001 (5.0 × 10^5 Neltependocel + Y-27632 100 µM) | AURN001 (1.0 × 10^6 Neltependocel + Y-27632 100 µM)
Number analyzed (Participants) | 21 | 18 | 19 | 19 | 20
change in ETDRS letters
  Week 4 | -28.7 (24.57) | -24.6 (33.16) | -27.8 (29.64) | -26.9 (25.04) | -16.9 (27.14)
  Month 2: number analyzed (Participants) | 6 | 6 | 7 | 8 | 10
  Month 2 | -17.2 (21.69) | -20.5 (37.31) | -26.6 (29.37) | -24.3 (27.63) | -12.1 (28.37)
  Month 3 | -19.6 (25.82) | -8.1 (40.76) | -10.6 (22.64) | -9.2 (27.96) | 0.2 (21.73)
  Month 4.5 | -21.2 (26.51) | -8.9 (39.80) | -11.6 (26.97) | -4.1 (28.07) | 5.4 (19.90)
  Month 6 | -21.2 (28.63) | -5.6 (40.48) | -15.2 (25.26) | -3.9 (28.30) | 6.8 (18.67)
  Month 9 | -21.4 (28.15) | -5.5 (41.19) | -13.1 (26.36) | -3.8 (28.54) | 8.2 (18.98)
  Month 12 | -21.5 (28.00) | -1.2 (40.29) | -14.3 (26.16) | -1.6 (30.30) | 8.8 (21.46)

6. Secondary Outcome: Change From Baseline in CCT at All Other Timepoints
Description: as for outcome 3
Time Frame: Baseline (Day 1) and at Weeks 1 and 4, Months 2, 3, 4.5, 6, 9, and 12
Population: Full Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | Y-27632 100 µM | Neltependocel (1.0 × 10^6) | AURN001 (2.5 × 10^5 Neltependocel + Y-27632 100 µM) | AURN001 (5.0 × 10^5 Neltependocel + Y-27632 100 µM) | AURN001 (1.0 × 10^6 Neltependocel + Y-27632 100 µM)
Number analyzed (Participants) | 21 | 18 | 19 | 19 | 20
Microns
  Week 1 | 87.4 (89.76) | 116.9 (134.59) | 93.4 (155.81) | 69.4 (86.47) | 117.0 (138.71)
  Week 4 | 97.5 (117.81) | 77.3 (102.40) | 35.1 (126.58) | 40.7 (57.74) | 66.0 (78.97)
  Month 2: number analyzed (Participants) | 6 | 6 | 7 | 8 | 10
  Month 2 | 63.7 (61.40) | 64.4 (100.38) | 47.9 (45.15) | 2.6 (45.88) | 36.9 (72.53)
  Month 3 | 60.8 (115.35) | -4.6 (114.97) | -16.1 (94.48) | -1.6 (76.72) | 20.8 (68.96)
  Month 4.5 | 66.9 (117.55) | 6.3 (113.65) | -25.0 (110.49) | -11.8 (76.22) | 6.8 (65.26)
  Month 6 | 65.7 (116.75) | -5.7 (112.03) | -20.2 (110.13) | -16.7 (66.35) | 2.6 (70.27)
  Month 9 | 64.8 (122.48) | -15.5 (112.88) | -21.0 (114.96) | -37.3 (74.17) | -21.7 (50.56)
  Month 12 | 63.0 (114.77) | -22.4 (107.81) | -19.1 (113.35) | -31.8 (68.25) | -7.6 (89.14)

7. Secondary Outcome: Percentage of Participants Achieving ≥10-letter Improvement in BCVA at All Timepoints - Observed Data
Description: as for outcome 4
Time Frame: At Week 4 and at Months 2, 3, 4.5, 6, 9 and 12
Population: Full Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Number; unit: percentage of participants
Arm/Group | Y-27632 100 µM | Neltependocel (1.0 × 10^6) | AURN001 (2.5 × 10^5 Neltependocel + Y-27632 100 µM) | AURN001 (5.0 × 10^5 Neltependocel + Y-27632 100 µM) | AURN001 (1.0 × 10^6 Neltependocel + Y-27632 100 µM)
Number analyzed (Participants) | 21 | 17 | 19 | 19 | 20
percentage of participants
  Week 4 | 4.8 | 11.8 | 15.8 | 5.3 | 10.0
  Month 2: number analyzed (Participants) | 6 | 6 | 7 | 8 | 10
  Month 2 | 0 | 16.7 | 14.3 | 12.5 | 40.0
  Month 3: number analyzed (Participants) | 15 | 17 | 17 | 19 | 19
  Month 3 | 6.7 | 47.1 | 11.8 | 31.6 | 31.6
  Month 4.5: number analyzed (Participants) | 12 | 14 | 14 | 17 | 19
  Month 4.5 | 16.7 | 50.0 | 21.4 | 35.3 | 52.6
  Month 6: number analyzed (Participants) | 6 | 14 | 12 | 16 | 19
  Month 6 | 50.0 | 57.1 | 16.7 | 43.8 | 57.9
  Month 9: number analyzed (Participants) | 3 | 12 | 8 | 13 | 18
  Month 9 | 33.3 | 83.3 | 37.5 | 53.8 | 77.8
  Month 12: number analyzed (Participants) | 3 | 12 | 7 | 12 | 17
  Month 12 | 33.3 | 83.3 | 42.9 | 66.7 | 82.4

ADVERSE EVENTS:
Time Frame: From first dose (Day 1) through Month 12
Description: Treatment emergent adverse events (TEAEs) and serious TEAEs were collected from Safety Analysis Set which comprised of all eligible participants who received any amount of study drug during intracameral injection.
Arm/Group | Y-27632 100 µM | Neltependocel 1.0 × 10^6 | AURN001 (2.5 × 10^5 Neltependocel + Y-27632 100 µM) | AURN001 (5.0 × 10^5 Neltependocel + Y-27632 100 µM) | AURN001 (1.0 × 10^6 Neltependocel + Y-27632 100 µM)
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/18 | 0/19 | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/21 | 1/18 | 0/19 | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 9/21 | 11/18 | 10/19 | 18/19 | 14/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Y-27632 100 µM (N=21) | Neltependocel 1.0 × 10^6 (N=18) | AURN001 (2.5 × 10^5 Neltependocel + Y-27632 100 µM) (N=19) | AURN001 (5.0 × 10^5 Neltependocel + Y-27632 100 µM) (N=19) | AURN001 (1.0 × 10^6 Neltependocel + Y-27632 100 µM) (N=20)
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Y-27632 100 µM (N=21) | Neltependocel 1.0 × 10^6 (N=18) | AURN001 (2.5 × 10^5 Neltependocel + Y-27632 100 µM) (N=19) | AURN001 (5.0 × 10^5 Neltependocel + Y-27632 100 µM) (N=19) | AURN001 (1.0 × 10^6 Neltependocel + Y-27632 100 µM) (N=20)
Ocular hypertension (Eye disorders) | 3 | 2 | 3 | 2 | 1
Conjunctival haemorrhage (Eye disorders) | 2 | 0 | 1 | 1 | 2
Corneal epithelium defect (Eye disorders) | 0 | 1 | 0 | 1 | 1
Eye pain (Eye disorders) | 1 | 0 | 1 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 2 | 0 | 2
Punctate keratitis (Eye disorders) | 1 | 0 | 0 | 1 | 0
Detached Descemet's membrane (Eye disorders) | 0 | 1 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 1 | 0 | 0
Iridocele (Eye disorders) | 0 | 0 | 0 | 0 | 1
Iridocyclitis (Eye disorders) | 0 | 0 | 0 | 0 | 1
Iris adhesions (Eye disorders) | 0 | 0 | 1 | 0 | 0
Keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 1
Posterior capsule opacification (Eye disorders) | 0 | 0 | 1 | 0 | 0
Retinal vein occlusion (Eye disorders) | 0 | 1 | 0 | 0 | 0
Chalazion (Eye disorders) | 0 | 1 | 0 | 0 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Burns second degree (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 3 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 3 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 2 | 0
Influenza (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Knee arthroplasty (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 1 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Macular oedema (Eye disorders) | 1 | 0 | 0 | 1 | 1
Corneal degeneration (Eye disorders) | 1 | 0 | 0 | 1 | 0
Epiretinal membrane (Eye disorders) | 0 | 0 | 0 | 2 | 0
Corneal oedema (Eye disorders) | 0 | 0 | 1 | 0 | 0
Endocrine ophthalmopathy (Eye disorders) | 0 | 0 | 0 | 0 | 2
Ulcerative keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Abdominal hernia repair (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
Rotator cuff repair (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2024-09-23): https://cdn.clinicaltrials.gov/large-docs/56/NCT06041256/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-14): https://cdn.clinicaltrials.gov/large-docs/56/NCT06041256/SAP_001.pdf